CLINICAL TRIAL: NCT00156598
Title: Cobalt, Chromium and Titanium Serum Concentrations in Patients With Metal-on-Metal vs. Metal on Polyethylene Total Hip Replacements
Brief Title: Metal Ion Serum Concentrations in Patients With Total Hip Replacements
Status: Terminated | Type: Observational
Why Stopped: Resident graduated; faculty mentor retired
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 045-0031-006
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Osteoarthritis
Keywords: metal ion concentration
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Other research studies have shown that the levels of metals in the blood are slightly increased after patients receive a total hip replacement. We want to learn whether these elevated levels are associated with any adverse effects. We hope this study will help us identify which type of patients have elevated levels of metal in their blood.

DETAILED DESCRIPTION:
It is suspected that the concentration of the metals chromium, cobalt and titanium in the blood will be higher in people with an all metal total hip prosthesis than in those with a plastic and metal prosthesis. To find out if this is true, we will test blood samples for the levels of metal in the blood and compare the values from 3 groups of people:

1. people with metal on metal hip replacements
2. loosening of a plastic and metal prosthesis and
3. evidence of osteoarthritis and are awaiting a total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

Group 1 - unilateral hip replacement with metal on metal prosthesis, well functioning.

Group 2 - loosening of plastic and metal prosthesis Group 3 - osteoarthritis of the hip and awaiting total hip replacement

Exclusion Criteria:

* renal dysfunction
* other types of metal implants or dental prostheses
* rheumatoid arthritis
* hip infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Local surgeon's patients who have had a hip implant.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2004-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorence Trick, MD, Principal Investigator — University of Texas Health Science Center Department of Orthopaedics